CLINICAL TRIAL: NCT04495257
Title: A Phase I Study of APX005M in Combination With Nivolumab and Ipilimumab in Treatment Naïve Patients With Advanced Melanoma or Renal Cell Carcinoma
Brief Title: A Study of APX005M in Combination With Nivolumab and Ipilimumab in Treatment Naïve Patients With Advanced Melanoma or Renal Cell Carcinoma (RCC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Apexigen America, Inc. (Industry)
Responsible Party: Principal Investigator, Harriet Kluger, Professor of Medicine (Medical Oncology), Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026830
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: Advanced Melanoma; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab; sotigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (DL1) (Experimental): DL1 will include ipilimumab at 1mg/kg and nivolumab at 3 mg/kg with APX005M of 0.1mg/kg for the induction phase. After 4 cycles, participants will be treated with 360mg of nivolumab and APX005M every 3 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: APX005M
- Dose Level 2 (DL2) (Experimental): DL2 will include ipilimumab at 1mg/kg and nivolumab at 3 mg/kg with APX005M of 0.3mg/kg for the induction phase. After 4 cycles we will treat with 360mg of nivolumab and APX005M every 3 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: APX005M

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3mg/kg intravenously (IV) every 3 weeks for the first 4 treatments and then will be given at 360mg every 3 weeks thereafter
Drug: Ipilimumab — Ipilimumab 1mg/kg intravenously (IV) every 3 weeks for a total of 4 treatments
Drug: APX005M — APX005M 0.3mg/kg intravenously (IV) every 3 weeks

SUMMARY:
This study is a Phase 1, open-label, single institution, dose escalation and dose expansion study to evaluate the efficacy, safety, and tolerability of APX005M in combination with nivolumab and ipilimumab in patients with advanced melanoma and RCC.

DETAILED DESCRIPTION:
This trial is a phase 1 study to evaluate the safety and tolerability of APX005M in combination with nivolumab and ipilimumab. The study will enroll patients with advanced solid tumors (melanoma, RCC) to determine the recommended phase II dosing (RP2D) of APX005M in combination with ipilimumab 1mg/kg and nivolumab 3 mg/kg (IPI1 NIVO3) every 3 weeks for four cycles followed by APX005M in combination with nivolumab 360mg every 3 weeks. APX005M will be administered at a dose of 0.1 mg/kg every 3 weeks in Dose Level 1 (DL1) and escalated to 0.3 mg/kg every 3 weeks in Dose Level 2 (DL2) (Table 1). The IPI1 NIVO3 regimen is approved for patients with metastatic RCC.

APX005M is a humanized IgG1 agonistic monoclonal antibody that binds CD40. Nivolumab is a humanized IgG4 monoclonal antibody directed against PD-1. Ipilimumab is a humanized IgG1κ monoclonal antibody directed against CTLA-4.

Primary Objective

* To assess the safety and tolerability of APX005M in combination with nivolumab and ipilimumab
* To determine the recommended RP2D of APX005M in combination with nivolumab and ipilimumab in patients with unresectable metastatic melanoma or renal cell carcinoma.

Secondary Objective

• Determine rate and pattern of AEs in patients treated with APX005M in combination with nivolumab and ipilimumab

ELIGIBILITY:
Inclusion Criteria:

* 1. At least 1 site of disease must be accessible to provide repeat biopsies for tumor tissue. The biopsy may be waived if not feasible upon discussion with the study PIs. This site may be a target lesion as long as it will not be rendered unmeasurable by the biopsy procedure.

  2. Age ≥18, able to understand and sign the informed consent form 3. ECOG performance status < 2 4. No prior systemic immune therapy for advanced (unresectable) disease. Prior targeted therapy is allowed. Adjuvant therapy is allowed provided that at least 6 months have lapsed from the last dose of an immune checkpoint inhibitor. Prior small molecule inhibitors must be discontinued within 2 weeks before starting study.

  5. Life expectancy of at least 6 months 6. A history of previously treated brain metastases is allowed, provided that they are stable for at least 4 weeks.

  7. Willingness to undergo tumor biopsy (if amenable) prior to initiation of therapy and on trial.

  8. Willingness to provide an archival specimen block, if available, for research 9. Normal organ function . 10. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  11. Female subjects of childbearing potential should be willing to use a highly effective contraception (hormonal or IUD) or be surgically sterile, or abstain from heterosexual activity for a period of at least 5 months after the last dose of study drug. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

  12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through at least 7 months after the last dose of study drug.

  13. Patients must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST v1.1 criteria. Tumor sites situated in a previously irradiated area, or in an area subjected to other loco-reginal therapy, are not considered measurable unless there has been demonstrated progression in the lesion.

  14. Prior focal radiotherapy is allowed. Radiation to pulmonary or intestinal sites must be completed at least 1 week prior to study Day 1. Radiation to the brain must be completed within 4 weeks prior to initiation of treatment. There is no time restriction prior to study Day 1 for patients who have received radiation to bone, soft tissue or other sites. No radiopharmaceuticals (strontium, samarium) within 8 weeks before first dose of study drug administration.

  15. Major surgery must be completed at least 2 weeks prior to the first dose of study drug administration and patients should have recovered. Wounds must be healed.

Exclusion Criteria:

* 1. Untreated brain metastases. 2. A patient who has had prior treatment with immune therapy for advanced disease. Prior immune checkpoint inhibitors as adjuvant therapy is allowed provided at least 6 months have lapsed from the last dose. Prior targeted therapy is allowed as long as 2 weeks have passed.

  3. Use of corticosteroids to control immune related adverse events at enrollment will not be allowed, and patients who previously required corticosteroids for symptom control must be off steroids for at least 2 weeks. Low-dose steroid use (≤10 mg of prednisone or equivalent) as corticosteroid replacement therapy for primary or secondary adrenal insufficiency is allowed.

  4. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to prior treatments with the exceptions such as alopecia listed in Table 2.

  5. History of grade 3-4 neurologic or cardiac toxicity or life-threatening liver toxicity poorly responsive to steroids with prior anti-PD-1/anti-PD-L1 therapy in the adjuvant setting.

  6. Presence of leptomeningeal disease. 7. Has active autoimmune disease unrelated to use of immune checkpoint inhibitors that has required systemic treatment in the past year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

  8. Pregnancy or breast feeding. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, ipilimumab or APX005M, breastfeeding must be discontinued if the mother is enrolled on this trial.

  9. Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.

  10. Either a concurrent condition (including medical illness, such as active infection requiring treatment with intravenous antibiotics or the presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or a medical condition that confounds the ability to interpret data from the study.

  11. Concurrent, active malignancies in addition to those being studied (other than cutaneous squamous cell carcinoma or basal cell carcinoma).

  12. Active (non-infectious) pneumonitis. 13. Has a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) acute or chronic infection.

  14. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

  15. History of myocardial infarction or unstable angina within 3 months prior to Cycle 1, Day 1.

  16. Prisoners, or subjects who are under compulsory detention 17. Open wounds and active skin infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | Up to 2 years
  The safety and tolerability of APX005M in combination with nivolumab and ipilimumab will be assessed by monitoring the of dose-limiting toxicities (DLTs) . This will be defined by both DLTs and any of the following AEs (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v5.0) which occur during the first 9 weeks of ipilimumab + nivolumab + APX005M administration that is not clearly due to a cause other than study medication. DLTs in this study do not include reversible grade 3-4 irAEs, that are acceptable and expected with treatment regimens containing ipilimumab and nivolumab, but do include severe, irreversible, non-endocrine adverse events
Recommended dose of APX005M | Up to 2 years
  This outcome will determine the recommended phase II dose (RP2D) of APX005M in combination with nivolumab and ipilimumab in patients with unresectable or metastatic melanoma or renal cell carcinoma (RCC). The RP2D will be defined as a triplet regimen that does not exceed a grade 3-4 irAE rate of approximately 55% or lead to a significant increase in dose limiting toxicities (DLTs) specific to an ipilimumab + nivolumab containing regimen, particularly those which are severe, irreversible, and non-endocrine related events.

SECONDARY OUTCOMES:
Adverse Events Rate | Up to 2 years
  The rate of AEs in patients treated with APX005M in combination with nivolumab and ipilimumab will be assessed.
Adverse Events Frequency | Up to 2 years
  The frequency of AE type in patients treated with APX005M in combination with nivolumab and ipilimumab will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Yale University; Sarah Weiss, MD, Principal Investigator — Yale University; Kelly Olino, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No